CLINICAL TRIAL: NCT02178098
Title: A Placebo-Controlled, Randomized, Double-Blind, Parallel Group Study to Evaluate the Efficacy and Safety of ETC-1002 in Patients With Hypercholesterolemia and Hypertension
Brief Title: Evaluation of ETC-1002 in Participants With Hypercholesterolemia and Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1002-014
Record Dates: First submitted 2014-06-16; First posted 2014-06-30 (Estimated); Results first posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Hypercholesterolemia; Hypertension
Keywords: LDL; Cholesterol
MeSH Terms: conditions — Hypercholesterolemia; Hypertension | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ETC-1002 (Experimental): ETC-1002 180 mg/day
  Interventions: Drug: ETC-1002
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ETC-1002 — ETC-1002 capsules taken once daily
  Arms: ETC-1002
Drug: Placebo — Placebo capsules taken once daily
  Arms: Placebo

SUMMARY:
This Phase 2 study will assess the efficacy and safety of ETC-1002 monotherapy versus placebo in participants with hypercholesterolemia and hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Mean 24-hour ambulatory SBP greater than or equal to 130 mmHg
* or- Mean 24-hour ambulatory DBP greater than or equal to 80 mmHg
* Fasting LDL-C between 100 and 220 mg/dL
* Fasting triglycerides less than 400 mg/dL
* Body mass index (BMI) between 18 and 45 kg/m2

Exclusion Criteria:

* Known or suspected secondary hypertension or history of malignant hypertension
* Taking more than two anti-hypertension medications at the first visit
* History or current clinically significant cardiovascular disease
* History or current type 1 diabetes or type 2 diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2015-05-22 (Actual); Study Completion 2015-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medpace Medical Monitor, Study Director — Medpace, Inc.
Locations (38):
- United States (38):
  - Birmingham, Alabama
  - Muscle Shoals, Alabama
  - Chandler, Arizona
  - Glendale, Arizona
  - Los Angeles, California
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Hialeah, Florida
  - Oviedo, Florida
  - Pembroke Pines, Florida
  - Port Orange, Florida
  - Meridian, Idaho
  - Chicago, Illinois
  - Gurnee, Illinois
  - Indianapolis, Indiana
  - Paducah, Kentucky
  - Auburn, Maine
  - Olive Branch, Mississippi
  - Butte, Montana
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Endwell, New York
  - Wilmington, North Carolina
  - Cincinnati, Ohio
  - Lyndhurst, Ohio
  - Willoughby Hills, Ohio
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Downingtown, Pennsylvania
  - Site 1, Mt. Pleasant, South Carolina
  - Site 2, Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Kenosha, Wisconsin
  - Madison, Wisconsin

REFERENCES:
- [Background] Ballantyne CM, Davidson MH, Macdougall DE, Bays HE, Dicarlo LA, Rosenberg NL, Margulies J, Newton RS. Efficacy and safety of a novel dual modulator of adenosine triphosphate-citrate lyase and adenosine monophosphate-activated protein kinase in patients with hypercholesterolemia: results of a multicenter, randomized, double-blind, placebo-controlled, parallel-group trial. J Am Coll Cardiol. 2013 Sep 24;62(13):1154-62. doi: 10.1016/j.jacc.2013.05.050. Epub 2013 Jun 13. PMID 23770179
- [Background] Gutierrez MJ, Rosenberg NL, Macdougall DE, Hanselman JC, Margulies JR, Strange P, Milad MA, McBride SJ, Newton RS. Efficacy and safety of ETC-1002, a novel investigational low-density lipoprotein-cholesterol-lowering therapy for the treatment of patients with hypercholesterolemia and type 2 diabetes mellitus. Arterioscler Thromb Vasc Biol. 2014 Mar;34(3):676-83. doi: 10.1161/ATVBAHA.113.302677. Epub 2014 Jan 2. PMID 24385236
- [Background] Pinkosky SL, Filippov S, Srivastava RA, Hanselman JC, Bradshaw CD, Hurley TR, Cramer CT, Spahr MA, Brant AF, Houghton JL, Baker C, Naples M, Adeli K, Newton RS. AMP-activated protein kinase and ATP-citrate lyase are two distinct molecular targets for ETC-1002, a novel small molecule regulator of lipid and carbohydrate metabolism. J Lipid Res. 2013 Jan;54(1):134-51. doi: 10.1194/jlr.M030528. Epub 2012 Nov 1. PMID 23118444
- [Background] Filippov S, Pinkosky SL, Lister RJ, Pawloski C, Hanselman JC, Cramer CT, Srivastava RAK, Hurley TR, Bradshaw CD, Spahr MA, Newton RS. ETC-1002 regulates immune response, leukocyte homing, and adipose tissue inflammation via LKB1-dependent activation of macrophage AMPK. J Lipid Res. 2013 Aug;54(8):2095-2108. doi: 10.1194/jlr.M035212. Epub 2013 May 24. PMID 23709692

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received matching oral placebo capsules taken once daily for 6 weeks.
- ETC-1002 180 mg: Participants received oral bempedoic acid 180 milligrams (mg) daily for 6 weeks.
Period: Overall Study
Arm/Group | Placebo | ETC-1002 180 mg
Started | 72 | 71
Completed | 67 | 59
Not Completed | 5 | 12
Not completed — Withdrawal by Subject | 0 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Sponsor Request | 1 | 0
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for members of the Safety Population, comprised of all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ETC-1002 180 mg | Total
Number analyzed (Participants) | 72 | 71 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (8.29) | 54.6 (8.41) | 55.6 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 26 | 61
  Male | 37 | 45 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 2 | 3
  Black or African American | 23 | 17 | 40
  White | 45 | 49 | 94
  More than one race | 1 | 2 | 3
  Unknown | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated Low-density Lipoprotein Cholesterol (LDL-C) to Week 6
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Week -1 and Week 0. Percent change from Baseline in LDL-C was analyzed using an analysis of covariance (ANCOVA) model with a term for treatment and Baseline value as a covariate. The Week 6 endpoint was the last available post-Baseline value. For the Week 6 endpoint, missing values at Week 6 were imputed using the last observation carried forward (LOCF) procedure, with only post-Baseline values carried forward. Modified Intent-to-Treat (mITT) Population is defined as all randomized participants who received at least 1 dose of study drug, had a Baseline assessment, and had at least 1 post-Baseline assessment, excluding any assessment taken more than 2 days after a dose of study drug
Time Frame: Baseline; 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 72 | 68
Percent Change | 3.16 (2.133) | -21.08 (2.196)
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = -24.24, 95% CI 2-sided [-30.33 to -18.15], Standard Error of Mean 3.080 — The least squares mean difference was calculated as the value for the ETC-1002 180 mg arm minus the value for the placebo arm

2. Secondary Outcome: Change From Baseline in Mean 24-hour Systolic Blood Pressure (SBP) to Week 6
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Baseline was defined as the last value prior to the first dose of study medication. Change from Baseline was calculated using an ANCOVA model with a term for treatment and Baseline value as a covariate. The Week 6 endpoint was the last available post-Baseline value.
Time Frame: Baseline; 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Groups:
- ETC-1002 180 mg: Participants received oral bempedoic acid 180 mg daily for 6 weeks.
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 69 | 64
millimeters of mercury (mmHg) | -0.64 (1.045) | -2.28 (1.085)
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p = 0.2808, ANCOVA; Least squares mean difference = -1.64, 95% CI 2-sided [-4.62 to 1.35], Standard Error of Mean 1.511 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in 24-hour Mean Diastolic Blood Pressure (DBP) to Week 6
Description: as for outcome 2
Time Frame: Baseline; 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 69 | 64
mmHg | -0.05 (0.760) | -1.10 (0.790)
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p = 0.3461, ANCOVA; Least squares mean difference = -1.05, 95% CI 2-sided [-3.25 to 1.15], Standard Error of Mean 1.111 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Mean Daytime SBP to Week 6
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Baseline was defined as the last value prior to the first dose of study medication. Change from Baseline was calculated using an ANCOVA model with a term for treatment and Baseline value as a covariate. Daytime measurements were defined as those taken from 7 AM to 10 PM (>7 AM and ≤10 PM). The Week 6 endpoint was the last available post-Baseline value.
Time Frame: Baseline; 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 69 | 64
mmHg | -0.35 (1.198) | -2.66 (1.245)
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p = 0.1852, ANCOVA; Least squares mean difference = -2.31, 95% CI 2-sided [-5.74 to 1.12], Standard Error of Mean 1.734 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline in Mean Daytime DBP to Week 6
Description: as for outcome 4
Time Frame: Baseline; 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 69 | 64
mmHg | -0.01 (0.856) | -1.47 (0.890)
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p = 0.2481, ANCOVA; Least squares mean difference = -1.45, 95% CI 2-sided [-3.93 to 1.03], Standard Error of Mean 1.253 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline in Mean Nighttime SBP to Week 6
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Baseline was defined as the last value prior to the first dose of study medication. Change from Baseline was calculated using an ANCOVA model with a term for treatment and Baseline value as a covariate. Nighttime measurements were defined as those taken from 10 PM to 7 AM (>10 PM and ≤7 AM). The Week 6 endpoint was the last available post-Baseline value.
Time Frame: Baseline; 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 69 | 64
mmHg | -1.18 (1.167) | -1.57 (1.212)
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p = 0.8181, ANCOVA; Least squares mean difference = -0.39, 95% CI 2-sided [-3.72 to 2.94], Standard Error of Mean 1.684 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in Mean Nighttime DBP to Week 6
Description: as for outcome 6
Time Frame: Baseline; 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 69 | 64
mmHg | -0.52 (0.879) | -0.33 (0.913)
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p = 0.8817, ANCOVA; Least squares mean difference = 0.19, 95% CI 2-sided [-2.33 to 2.71], Standard Error of Mean 1.274 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline in Sitting Cuff SBP to Week 6
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Baseline was defined as the mean of the values from Weeks -1 and 0. Change from Baseline was calculated using an ANCOVA model with a term for treatment and Baseline value as a covariate. Three BP measurements were collected at least 3 minutes apart, and the mean of the second and third measurements was calculated and used for summary and analysis. The Week 6 endpoint was the last available post-Baseline value.
Time Frame: Baseline: 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 72 | 68
mmHg | -4.98 (1.274) | -3.45 (1.311)
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p = 0.4040, ANCOVA; Least squares mean difference = 1.53, 95% CI 2-sided [-2.09 to 5.15], Standard Error of Mean 1.829 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change From Baseline in Sitting Cuff DBP to Week 6
Description: as for outcome 8
Time Frame: Baseline; 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 72 | 68
mmHg | -3.32 (0.820) | -2.53 (0.844)
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p = 0.5061, ANCOVA; Least squares mean difference = 0.79, 95% CI 2-sided [-1.54 to 3.11], Standard Error of Mean 1.178 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Percent Change From Baseline in High-sensitivity C-reactive Protein (hsCRP) to Week 6
Description: A non-parametric analysis was performed for hsCRP parameters. Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the last value prior to the first dose of study medication. If hsCRP was <0.2, 0.1 was imputed for analysis. The Week 6 endpoint was the last available post-Baseline value.
Time Frame: Baseline; 6 weeks
Population: miTT Population. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 69 | 61
Percent Change | 19.61 [-16.67 to 64.29] | -25.00 [-50.85 to 0.00]
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p < 0.0001, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = -43.64, 95% CI 2-sided [-62.80 to -25.21] — The 95% confidence interval (CI) was calculated using Hodges-Lehmann analysis

11. Secondary Outcome: Percent Change From Baseline in Total Cholesterol to Week 6
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Week -1 and Week 0. Change from Baseline was calculated using an ANCOVA model with terms for treatment and statin intolerance, and value as a covariate. The Week 6 endpoint was the last available post-Baseline value.
Time Frame: Baseline; 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 72 | 68
Percent Change | 2.90 (1.389) | -13.77 (1.430)
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = -16.67, 95% CI 2-sided [-20.63 to -12.70], Standard Error of Mean 2.006 — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (ApoB) to Week 6
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Week -1 and Week 0. Change from Baseline was calculated using an ANCOVA model with terms for treatment and statin intolerance, and Baseline value as a covariate. The Week 6 endpoint was the last available post-Baseline value.
Time Frame: Baseline; 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 69 | 61
Percent Change | 4.77 (1.797) | -14.13 (1.911)
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = -18.90, 95% CI 2-sided [-24.09 to -13.71], Standard Error of Mean 2.624 — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Percent Change From Baseline in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) to Week 6
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the last value prior to the first dose of study medication. Change from Baseline was calculated using an ANCOVA model with a term for treatment and Baseline value as a covariate. The Week 6 endpoint was the last available post-Baseline value.
Time Frame: Baseline; 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 72 | 68
Percent Change | 3.20 (1.728) | -15.49 (1.779)
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = -18.69, 95% CI 2-sided [-23.62 to -13.77], Standard Error of Mean 2.490 — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG) to Week 6
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Week -1 and Week 0. The Week 6 endpoint was the last available post-Baseline value. Data was analyzed using non-parametric analysis.
Time Frame: Baseline; 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 72 | 68
Percent Change | -3.75 [-18.67 to 15.69] | -0.07 [-20.63 to 36.38]
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p = 0.3689, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 5.25, 95% CI 2-sided [-6.78 to 16.42] — The 95% CI was calculated using Hodges-Lehmann analysis

15. Secondary Outcome: Percent Change From Baseline in HDL-C to Week 6
Description: as for outcome 12
Time Frame: Baseline; 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 72 | 68
Percent Change | 2.42 (1.614) | -5.76 (1.661)
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p = 0.0006, ANCOVA; Least squares mean difference = -8.18, 95% CI 2-sided [-12.76 to -3.59], Standard Error of Mean 2.319 — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Percent Change From Baseline in Free Fatty Acids (FFA) to Week 6
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Week -1 and Week 0. The Week 6 endpoint was the last available post-Baseline value.
Time Frame: Baseline; 6 weeks
Population: mITT Population. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 68 | 61
Percent Change | 1.08 [-23.81 to 30.46] | 9.56 [-19.49 to 43.53]
Statistical Analysis 1: Comparison: Placebo vs ETC-1002 180 mg; Test type: Superiority; p = 0.3093, Wilcoxon Rank-Sum Test; Median Difference (Final Values) = 7.60, 95% CI 2-sided [-8.21 to 24.02] — The 95% CI was calculated using Hodges-Lehmann analysis

17. Secondary Outcome: Change From Baseline in Body Weight to Week 6
Description: Baseline was defined as the mean of the values from Week -1 and Week 0. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; 6 weeks
Population: Safety Population: all randomized participants who received at least 1 dose of study drug. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo | ETC-1002 180 mg
Number analyzed (Participants) | 67 | 57
kilograms | -0.335 (1.590) | -0.009 (1.927)

18. Secondary Outcome: Plasma Trough Concentrations of ETC-1002 and Metabolite ESP15228
Description: Plasma trough concentration is defined as the lowest concentration reached before the next dose is administered.
Time Frame: Week 2, Week 4 and Week 6
Population: Pharmacokinetic Concentration Population: all randomized participants who received at least 1 dose of study drug and had at least 1 measurable plasma concentration value for study drug collected between 18 and 36 hours post-dose. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | ETC-1002 180 mg
Number analyzed (Participants) | 70
nanograms per milliliter (ng/mL)
  Week 2, ETC-1002: number analyzed (Participants) | 64
  Week 2, ETC-1002 | 6666.20 (4777.661)
  Week 4, ETC-1002: number analyzed (Participants) | 60
  Week 4, ETC-1002 | 6817.45 (4543.944)
  Week 6, ETC-1002: number analyzed (Participants) | 58
  Week 6, ETC-1002 | 6836.36 (3702.241)
  Week 2, ESP15228: number analyzed (Participants) | 64
  Week 2, ESP15228 | 1219.60 (783.00)
  Week 4, ESP15228: number analyzed (Participants) | 60
  Week 4, ESP15228 | 1220.79 (674.437)
  Week 6, ESP15228: number analyzed (Participants) | 58
  Week 6, ESP15228 | 1221.32 (557.930)

ADVERSE EVENTS:
Time Frame: Up to approximately 14 weeks
Description: The analysis was performed using the Safety Population, which comprised of all randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo | ETC-1002 180 mg
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/71
Serious Adverse Events (participants affected / at risk) | 2/72 | 4/71
Other Adverse Events (participants affected / at risk) | 4/72 | 3/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | ETC-1002 180 mg (N=71)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | ETC-1002 180 mg (N=71)
Headache (Nervous system disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Principal Investigator plans to publish information from the study, a copy of the manuscript should be provided to the Sponsor for review before submission for publication or presentation. The Sponsor may request that the publication be withheld.